CLINICAL TRIAL: NCT06841315
Title: A Phase 1, Open-Label, Single-Dose Study to Evaluate the Pharmacokinetics, Safety, and Tolerability of Varegacestat in Participants With or Without Hepatic Impairment
Brief Title: A Varegacestat Hepatic Impairment Study
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Immunome, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: AL102-503
Record Dates: First submitted 2025-01-24; First posted 2025-02-24 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2026-01

CONDITIONS: Healthy Volunteer; Hepatic Impairment (HI)

STUDY DESIGN:
Intervention Model Description: Healthy participants (Group 1) will be matched by age (± 10 years), body mass index (BMI, ± 15%), and sex to participants with mild to moderate hepatic impairment (Groups 2 and 3). Participants with severe hepatic impairment (Group 4) will be included as needed and matched to Group 1.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment Arm (Experimental): Single oral dose of varegacestat administered on study day 1
  Interventions: Drug: varegacestat

INTERVENTIONS:
Drug: varegacestat — experimental intervention

SUMMARY:
This clinical trial is designed to determine the pharmacokinetics, safety and tolerability of varegacestat in people with impaired liver function compared to people with normal liver function.

DETAILED DESCRIPTION:
This is an open-label, single-dose, parallel study to evaluate the effects of varying degrees of impaired hepatic function on the PK, safety, and tolerability of varegacestat in adult participants.

The study will be conducted sequentially. The study will enroll participants with mild (Group 2) and moderate (Group 3) hepatic impairment (HI) and healthy participants with normal hepatic function (Group 1) at a 1:1 ratio. Matched healthy participants may match to more than one participant in the HI groups. Subsequently, if appropriate, the study will enroll participants with severe (Group 4) HI and healthy participants with normal hepatic function (Group 1), as needed, to provide 1:1 matches for Group 4. The decision to conduct Group 4 enrollment will be contingent upon the assessment of the feasibility, PK, and safety data from Groups 1-3.

ELIGIBILITY:
Inclusion Criteria (Healthy Participants):

* Healthy, adult, male or female (of nonchildbearing potential only), 18 to 84 years of age, inclusive, at the screening visit. Participant will be matched by age (± 10 years) and sex to a participant with hepatic impairment (HI). Each healthy participant may be matched to more than 1 participant with HI, but cannot be matched to more than 1 participant within the same HI group.
* Medically healthy with no clinically significant medical history, physical examination, clinical laboratory profiles, vital signs, and ECGs as deemed by the PI or designee

Inclusion Criteria (Hepatic Impairment):

* Healthy, apart from HI, adult male or female (of nonchildbearing potential only), 18 to 84 years of age, inclusive, at the screening visit.
* Considered to have HI (of any etiology) that has been clinically stable (no acute episodes of illness due to deterioration in hepatic function) for at least 1 month prior to dosing per the PI and Sponsor and is likely to remain stable throughout the study. To be classified as having hepatic impairment with known medical history of liver disease (with or without a known history of alcohol abuse).
* Has a score on the Child-Pugh scale at screening visit and confirmed at check-in as follows:

Mild: ≥5 and ≤6 [Category A]; or

Moderate: ≥7 and ≤9 [Category B]; or

Severe: ≥10 and ≤15 [Category C].

- Medically healthy, apart from HI, with no clinically significant medical history, physical examination, clinical laboratory profiles, vital signs, and ECGs as deemed by the PI or designee

Exclusion Criteria (Healthy Volunteers):

* Is mentally or legally incapacitated or has significant emotional problems at the time of the screening visit or expected during the conduct of the study.
* History or presence of clinically significant medical or psychiatric condition or disease in the opinion of the PI or designee.
* History of any illness that, in the opinion of the PI or designee, might confound the results of the study or pose an additional risk to the participant by their participation in the study.

Exclusion Criteria (Hepatic Impairment):

Participants must not be enrolled in the study, if they meet any of the following criteria:

* Is mentally or legally incapacitated or has significant emotional problems at the time of the screening visit or expected during the conduct of the study.
* History or presence of clinically significant medical (except for HI) or psychiatric condition or disease in the opinion of the PI or designee.
* History of any illness that, in the opinion of the PI or designee, might confound the results of the study or pose an additional risk to the participant by their participation in the study.

Ages: 18 Years to 84 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 44 (Estimated)
Dates: Start 2025-03-07 (Actual); Primary Completion 2025-11-05 (Actual); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
PK of varegacestat and metabolite from a single oral dose of varegacestat in hepatic impaired adult participants to matched healthy adult participants. | Up to 4 weeks
  AUC0-t varegacestat and metabolite
PK of varegacestat and metabolite from a single oral dose of varegacestat in hepatic impaired adult participants to matched healthy adult participants. | Up to 4 weeks
  AUC0-inf for varegacestat and metabolite
PK of varegacestat and metabolite from a single oral dose of varegacestat in hepatic impaired adult participants to matched healthy adult participants. | Up to 4 weeks
  Cmax for varegacestat and metabolite

SECONDARY OUTCOMES:
Assess the safety and tolerability of a single oral dose of varegacestat in hepatic impaired adult participants and in matched healthy adult participants. | Up to 4 weeks
  Number of subjects who experience treatment emergent adverse events (TEAEs)
Assess the safety and tolerability of a single oral dose of varegacestat in hepatic impaired adult participants and in matched healthy adult participants. | Up to 4 weeks
  Number of subjects who experience abnormalities in vital signs and in clinical laboratory tests such as serum chemistry and hematology
Assess the safety and tolerability of a single oral dose of varegacestat in hepatic impaired adult participants and in matched healthy adult participants. | Up to 4 weeks
  Number of subjects who experience 12-lead ECG abnormalities

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Orlando Clinical Research Center, Orlando, Florida
  - The Texas Liver Institute, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: Undecided